CLINICAL TRIAL: NCT02829008
Title: A Phase 2 Clinical Trial:Low -Dose-bevacizumab and Pemetrexed Versus Treatment of Physician's Choice in Metastatic HER2-negative Breast Cancer Patients After Failure of Taxanes and Anthracycline-containing Regimens
Brief Title: Low -Dose-bevacizumab and Pemetrexed Versus TPC in Metastatic HER2-negative Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LQ002; CAMS-LQOO2 (Other: CAMS)
Record Dates: First submitted 2016-07-03; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2 negative breast cancer; low-dose bevacizumab; pemetrexed
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low-dose-bevacizumab/Pemetrexed (Experimental): Low-dose-bevacizumab is given at a dose of 2 mg/kg once weekly by intravenous transfusion, which is on day 1, 8 and 15, and every three weeks are a treatment cycle .Pemetrexed is given at a dose of 500mg/m2 once on the first day by intravenous transfusion, and repeated every three weeks, too. The pretreatment of pemetrexed should be conducted within the study.
  Interventions: Drug: low-dose-bevacizumab/pemetrexed
- Treatment of physician' choice (Active Comparator): Treatment of physician's choice can be any drug or regimen that has been approved in metastatic cancer at present, including monotherapy, combination therapy, target therapy and palliative therapy. It can be drugs like taxanes,capecitabine, gemcitabine, cisplatin, everolimus or even nutrient solution,et al.
  Interventions: Drug: Treatment of physician's choice

INTERVENTIONS:
Drug: low-dose-bevacizumab/pemetrexed — Bevacizumab is administrated at a dose of 2 mg/kg once weekly by intravenous transfusion, which is on day 1, 8 and 15, and pemetrexed is given at a dose of 500mg/m2 once on the first day by intravenous transfusion, and repeated every three weeks, too.
  Other Names: Avastin/ALIMTA
  Arms: low-dose-bevacizumab/Pemetrexed
Drug: Treatment of physician's choice — The clinicians can select any drug or regimen that has been approved in metastatic cancer at present, including monotherapy, combination therapy, target therapy and palliative therapy. Specific agents include taxanes, capecitabine, gemcitabine, vinorelbine, cisplatin,carboplatin, nutrient solutions, and so on. These agents can be administered as monotherapy or in combination.
  Other Names: any drug or regimen approved in metastatic cancer
  Arms: Treatment of physician' choice

SUMMARY:
This is a single-center, open, randomized, controlled phase 2 clinical trial designed to compare low-dose-bevacizumab and pemetrexed with TPC in metastatic HER2-negative breast cancer patients after failure of taxanes and anthracycline-containing regimens.

DETAILED DESCRIPTION:
There is no standard therapy for advanced human epidermal growth factor receptor 2 (HER2) -negative breast cancer patients after failure of taxanes and anthracycline-containing regimens at present. Pemetrexed is a multitargeted antimetabolite. Its efficacy in metastatic breast cancer has been confirmed in several small sample size studies and meta-analyses. Its response rate (RR) is about 30%, and will be higher in HER2-negative breast cancer. However, there is no study focused on this subtype of breast cancer. Bevacizumab is also an effective alternative for metastatic breast cancer. Several studies indicate that the combination of bevacizumab and chemotherapy could improve both RR and overall survival, but its use is confined by its severe side effect and far from adequate treatment. Recent years, a lot of studies have assessed the efficacy of metronomic chemotherapy. Metronomic therapy refers to the chronic administration of low doses of cytotoxic drugs at close, regular intervals. It could promote the apoptosis of tumor endothelial cell , continuously inhibit tumor angiogenesis, and exhibit a significant superiority of low toxicity, reduced cost and prolonged combination therapy period. According to reports in literature, the expression of anti-angiogenic biomarkers, such as,vascular endothelial growth factor(VEGF)-A, VEGF-C, soluble vascular endothelial growth factor receptor (sVEGFR)-1, sVEGFR-2,thrombospondin-1(TSP-1), platelet factor 4 (PF-4) might be concerned with the efficacy of metronomic therapy. Since there are no reported clinical trials according to metronomic bevacizumab in HER2-negative breast cancer, the investigators come up with this study. In this study, the investigators try to make a comparison of the efficacy and safety of low-dose-bevacizumab and pemetrexed with treatment of physician's choice (TPC) in metastatic breast cancer after failure of taxanes and anthracycline-containing regimens, to validate the correlative biomarkers and to find an optimal choice for previously treated metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic breast cancer females confirmed by pathological and/or cytological examination;
2. Breast cancer patients who received taxanes and anthracycline-containing regimens previously;
3. HER2-negative breast cancer patients confirmed by immunohistochemical test or fluorescent in situ hybridization(FISH);
4. Patients aged from 18-70 years old, and patients with Eastern Cooperative Oncology Group（ECOG） performance status scored 0-2;
5. One or more measurable lesions in imaging examination,with a diameter no less than 20mm in ordinary computed tomography (CT) or magnetic resonance imaging (MRI), or a scanning diameter no less than 10mm in spiral CT;
6. Any other kind of concomitant chemotherapy is not allowed during the research. If the patients had accepted other chemotherapy before recruitment, he can enter into the study until the drug is eliminated 30 days later;
7. Patients without any kind of major organ dysfunction: normal blood test results, normal function of heart, liver, kidney, marrow and so on.

Exclusion Criteria:

1. Patients who had received any chemotherapy, radiotherapy, biotherapy, or drugs and physical treatment in other clinical trials four weeks within the enrollment;
2. Patients who has no measurable or assessable lesions ;
3. Patients with moderate or severe liver dysfunction
4. Pregnant or lactational patients;
5. Patients with severe complications, including severe heart disease, cerebrovascular disease, uncontrolled diabet and hypertension, severe infection , active peptic ulcer and so on;
6. Patient who had previously received pemetrexed-containing regimens in metastatic setting.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rare (ORR) | up to 24 months
  Evaluated as complete remission(CR) and partial remission(PR) according to Response Evaluation Criteria in Solid Tumors (RECIST)version 1.1

SECONDARY OUTCOMES:
progression free survival(PFS) | up to 48 months
Overall survival(OS) | up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD., Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bauer KR, Brown M, Cress RD, Parise CA, Caggiano V. Descriptive analysis of estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and HER2-negative invasive breast cancer, the so-called triple-negative phenotype: a population-based study from the California cancer Registry. Cancer. 2007 May 1;109(9):1721-8. doi: 10.1002/cncr.22618. PMID 17387718
- [Background] Kassam F, Enright K, Dent R, Dranitsaris G, Myers J, Flynn C, Fralick M, Kumar R, Clemons M. Survival outcomes for patients with metastatic triple-negative breast cancer: implications for clinical practice and trial design. Clin Breast Cancer. 2009 Feb;9(1):29-33. doi: 10.3816/CBC.2009.n.005. PMID 19299237
- [Background] Isakoff SJ, Mayer EL, He L, Traina TA, Carey LA, Krag KJ, Rugo HS, Liu MC, Stearns V, Come SE, Timms KM, Hartman AR, Borger DR, Finkelstein DM, Garber JE, Ryan PD, Winer EP, Goss PE, Ellisen LW. TBCRC009: A Multicenter Phase II Clinical Trial of Platinum Monotherapy With Biomarker Assessment in Metastatic Triple-Negative Breast Cancer. J Clin Oncol. 2015 Jun 10;33(17):1902-9. doi: 10.1200/JCO.2014.57.6660. Epub 2015 Apr 6. PMID 25847936
- [Background] Robert NJ, Conkling PR, O'Rourke MA, Kuefler PR, McIntyre KJ, Zhan F, Asmar L, Wang Y, Shonukan OO, O'Shaughnessy JA. Results of a phase II study of pemetrexed as first-line chemotherapy in patients with advanced or metastatic breast cancer. Breast Cancer Res Treat. 2011 Feb;126(1):101-8. doi: 10.1007/s10549-010-1286-0. Epub 2010 Dec 25. PMID 21188632
- [Background] Martin M. Clinical Experience With Pemetrexed in Breast Cancer. Semin Oncol. 2006 Feb;33(Suppl 2):S15-8. doi: 10.1053/j.seminoncol.2005.07.027. PMID 16472713
- [Background] Garin A, Manikhas A, Biakhov M, Chezhin M, Ivanchenko T, Krejcy K, Karaseva V, Tjulandin S. A phase II study of pemetrexed and carboplatin in patients with locally advanced or metastatic breast cancer. Breast Cancer Res Treat. 2008 Jul;110(2):309-15. doi: 10.1007/s10549-007-9722-5. Epub 2007 Sep 13. PMID 17851759
- [Background] Miller K, Wang M, Gralow J, Dickler M, Cobleigh M, Perez EA, Shenkier T, Cella D, Davidson NE. Paclitaxel plus bevacizumab versus paclitaxel alone for metastatic breast cancer. N Engl J Med. 2007 Dec 27;357(26):2666-76. doi: 10.1056/NEJMoa072113. PMID 18160686
- [Background] Miles DW, Chan A, Dirix LY, Cortes J, Pivot X, Tomczak P, Delozier T, Sohn JH, Provencher L, Puglisi F, Harbeck N, Steger GG, Schneeweiss A, Wardley AM, Chlistalla A, Romieu G. Phase III study of bevacizumab plus docetaxel compared with placebo plus docetaxel for the first-line treatment of human epidermal growth factor receptor 2-negative metastatic breast cancer. J Clin Oncol. 2010 Jul 10;28(20):3239-47. doi: 10.1200/JCO.2008.21.6457. Epub 2010 May 24. PMID 20498403
- [Background] Robert NJ, Dieras V, Glaspy J, Brufsky AM, Bondarenko I, Lipatov ON, Perez EA, Yardley DA, Chan SY, Zhou X, Phan SC, O'Shaughnessy J. RIBBON-1: randomized, double-blind, placebo-controlled, phase III trial of chemotherapy with or without bevacizumab for first-line treatment of human epidermal growth factor receptor 2-negative, locally recurrent or metastatic breast cancer. J Clin Oncol. 2011 Apr 1;29(10):1252-60. doi: 10.1200/JCO.2010.28.0982. Epub 2011 Mar 7. PMID 21383283
- [Background] Browder T, Butterfield CE, Kraling BM, Shi B, Marshall B, O'Reilly MS, Folkman J. Antiangiogenic scheduling of chemotherapy improves efficacy against experimental drug-resistant cancer. Cancer Res. 2000 Apr 1;60(7):1878-86. PMID 10766175
- [Background] Kerbel RS, Kamen BA. The anti-angiogenic basis of metronomic chemotherapy. Nat Rev Cancer. 2004 Jun;4(6):423-36. doi: 10.1038/nrc1369. No abstract available. PMID 15170445
- [Background] Wong NS, Buckman RA, Clemons M, Verma S, Dent S, Trudeau ME, Roche K, Ebos J, Kerbel R, Deboer GE, Sutherland DJ, Emmenegger U, Slingerland J, Gardner S, Pritchard KI. Phase I/II trial of metronomic chemotherapy with daily dalteparin and cyclophosphamide, twice-weekly methotrexate, and daily prednisone as therapy for metastatic breast cancer using vascular endothelial growth factor and soluble vascular endothelial growth factor receptor levels as markers of response. J Clin Oncol. 2010 Feb 10;28(5):723-30. doi: 10.1200/JCO.2009.24.0143. Epub 2009 Dec 21. PMID 20026801
- [Background] Mayer EL, Isakoff SJ, Klement G, Downing SR, Chen WY, Hannagan K, Gelman R, Winer EP, Burstein HJ. Combination antiangiogenic therapy in advanced breast cancer: a phase 1 trial of vandetanib, a VEGFR inhibitor, and metronomic chemotherapy, with correlative platelet proteomics. Breast Cancer Res Treat. 2012 Nov;136(1):169-78. doi: 10.1007/s10549-012-2256-5. Epub 2012 Sep 23. PMID 23001754
- [Background] Perroud HA, Rico MJ, Alasino CM, Pezzotto SM, Rozados VR, Scharovsky OG. Association between baseline VEGF/sVEGFR-2 and VEGF/TSP-1 ratios and response to metronomic chemotherapy using cyclophosphamide and celecoxib in patients with advanced breast cancer. Indian J Cancer. 2013 Apr-Jun;50(2):115-21. doi: 10.4103/0019-509X.117031. PMID 23979202
- [Background] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385